CLINICAL TRIAL: NCT05136287
Title: SEMAGLUTIDE VERSUS GLP-1 RECEPTOR AGONISTS. EFFECTIVENESS , SAFETY AND QUALITY OF LIFE IN PATIENTS WITH DIABETES MELLITUS 2. OBSERVATIONAL, PROSPECTIVE AND MULTICENTER STUDY. SEVERAL STUDY.
Acronym: SEVERAL
Status: Completed | Type: Observational
Sponsor: Jose Seijas Amigo (Other)
Responsible Party: Sponsor-Investigator, Jose Seijas Amigo, Principal Investigator, Hospital Clinico Universitario de Santiago
Organization: Hospital Clinico Universitario de Santiago (Other)
Other Study IDs: SEVERAL
Record Dates: First submitted 2021-11-12; First posted 2021-11-29 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Weight Loss; Diabetes Mellitus, Type 2; Quality of Life; Safety Issues
Keywords: semaglutide; GLP1 receptor agonists; diabetes mellitus 2; weight loss; BMI
MeSH Terms: conditions — Weight Loss; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diabetes mellitus 2 patients with obesity: Patients that meet criteria to start treatment with GLP-1 receptor agonists (dulaglutide; exenatide; liraglutide; lixisenatide )
  Interventions: Drug: GLP-1 receptor agonist

INTERVENTIONS:
Drug: GLP-1 receptor agonist — Patients are included after GLP1 agonists prescription , at the first dispensation

SUMMARY:
Introduction:

GLP-1 receptor agonists (aGLP1) act increasing pancreatic insulin secretion in response to the glucose, they reduce glucagon secretion and reduce appetite by acting in the central level. Several aGLP1 were approved through different clinical trials where they showed efficacy in the glycemic control and reduction in cardiovascular events. They also showed weight loss in different clinical trials with patients with diabetes mellitus 2 (DM2) and also in specific clinical trial where the weight loss was the primary endpoint (STEP study).

Objective:

The objective is to evaluate and compare the weight loss in patients with DM2 treated with the different aGLP1 for the first time. Secondary endpoints are HbA1c reduction, changes in quality of life and physical activity and the safety of these drugs.

Design:

It is a postauthorization, multicenter, non-randomized and prospective study. Patients that will start treatment for the first time with aGLP1 will be recruited in 10 primary care centers in SERGAS Galician Hospitals for a period of 6 months and 44 weeks of follow-up. The primary endpoint will be to evaluate the wight loss with the different aGLP1 and the secondary endpoint will be HbA1c reduction, changes in the quality of life through the EuroQol-5D and changes physical activity through the SF-12 questionnaire, and also the safety of these drugs. The sample size will be of 360 patients.

Statistical analysis:

Previous studies showed efficacy in weight loss with semaglutide about (3,6-4,9 kg), while with other aGLP1 the weight loss was smaller , about (0,86-2,96 kg).

Based in these data and with a 5% of significance level, a weight loss average in the aGLP1 group of 2,5 kg, average in semaglutide group of 4,2 kg, and combination deviation of 3,0kg, including 360 subjects we will have a statistical power above 90% to detect differences through T-test for independent samples.

The justification of this simple size was performed with the statistical software SPSS 3.0

Conclusions:

The SEVERAL study will try to provide information about weight loss efficacy, changes in quality of life, physical activity and safety of the aGLP1in patients with DM2 that start treatment with these drugs in the real life (Real-World Evidence)

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or over
* To start with the first funded dose of GLP1 receptor agonists ( BMI > 30Kg/m2)
* Treated with another oral antidiabetic

Exclusion Criteria:

* Diagnosis of diabetic retinopahty and family history of thyroid cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Diabetes mellitus 2 with another oral antidibetic and obesity (BMI > 30Kg/m2) that present uncontrolled HbA1c. With a first prescription of GLP-1 receptor agonists.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Weight loss | 11 months
  The primary outcome will be by assesment of % weight loss
Weight loss | 11 months
  Assesment the weiht loss by reduction in Kg
Weight loss | 11 months
  Assesment of changes in BMI ( weight (Kg) and height (cm) will be combined to report BMI in kg/m^2)

SECONDARY OUTCOMES:
HbA1c values | 11 months
  HbA1c changes will be assessed during the study by routine sample tests (%)
Changes in Quality of life | 11 months
  By using the questionnaire called EuroQol EQ-5D-3L assessment. It has 2 parts, the first one has 5 questions with 3 possible answers (5 dimensions and 3 levels), so each health status has a rate called EVA from 1,0000 (the highest value) to - 0,5095 (the worst health status).
  The second part is a visual self-assessment between 0 (the worst health status) and 100 (the best health status). https://euroqol.org/
Changes in Physical Activity | 11 months
  By using the questionnaire called EuroQol SF-12 assessment.For each of the 8 dimensions, the items are coded, added and transformed on a scale that ranges from 0 (the worst health status for that dimension) to 100 (the best health status).
Number of participants experiencing adverse events | 11 months
  Gastrointestinal events; hypoglycemia; pancreatitis; fatigue; ijection reactions; Diabetic retinopathy; cardiac events and other possible events

CONTACTS AND LOCATIONS:
Overall Officials: Jose Seijas Amigo, Study Chair — Hospital Clínico Santiago de Compostela
Locations (11):
- Spain (11):
  - Centro de Salud de Culleredo, Culleredo, A Coruña
  - Centro de Salud de Fene, Fene, A Coruña
  - Centro de Salud de Ribeira, Ribeira, A Coruña
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Centro de Salud de Ribadeo, Ribadeo, Lugo
  - Centro de Salud de Vilalba, Vilalba, Lugo
  - Centro de Salud de O Carballiño, O Carballiño, Ourense
  - Centro de Salud Valmiñor, Nigrán, Pontevedra
  - Centro de Salud de O Ventorrillo, A Coruña
  - Centro de Salud de San Roque, Lugo
  - Centro de Salud Virxe Peregrina, Pontevedra

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] DeFronzo RA, Eldor R, Abdul-Ghani M. Pathophysiologic approach to therapy in patients with newly diagnosed type 2 diabetes. Diabetes Care. 2013 Aug;36 Suppl 2(Suppl 2):S127-38. doi: 10.2337/dcS13-2011. No abstract available. PMID 23882037
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Emerging Risk Factors Collaboration; Sarwar N, Gao P, Seshasai SR, Gobin R, Kaptoge S, Di Angelantonio E, Ingelsson E, Lawlor DA, Selvin E, Stampfer M, Stehouwer CD, Lewington S, Pennells L, Thompson A, Sattar N, White IR, Ray KK, Danesh J. Diabetes mellitus, fasting blood glucose concentration, and risk of vascular disease: a collaborative meta-analysis of 102 prospective studies. Lancet. 2010 Jun 26;375(9733):2215-22. doi: 10.1016/S0140-6736(10)60484-9. PMID 20609967
- [Background] Verspohl EJ. Novel therapeutics for type 2 diabetes: incretin hormone mimetics (glucagon-like peptide-1 receptor agonists) and dipeptidyl peptidase-4 inhibitors. Pharmacol Ther. 2009 Oct;124(1):113-38. doi: 10.1016/j.pharmthera.2009.06.002. Epub 2009 Jun 21. PMID 19545590
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Background] Marso SP, Daniels GH, Brown-Frandsen K, Kristensen P, Mann JF, Nauck MA, Nissen SE, Pocock S, Poulter NR, Ravn LS, Steinberg WM, Stockner M, Zinman B, Bergenstal RM, Buse JB; LEADER Steering Committee; LEADER Trial Investigators. Liraglutide and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):311-22. doi: 10.1056/NEJMoa1603827. Epub 2016 Jun 13. PMID 27295427
- [Background] Gerstein HC, Colhoun HM, Dagenais GR, Diaz R, Lakshmanan M, Pais P, Probstfield J, Riesmeyer JS, Riddle MC, Ryden L, Xavier D, Atisso CM, Dyal L, Hall S, Rao-Melacini P, Wong G, Avezum A, Basile J, Chung N, Conget I, Cushman WC, Franek E, Hancu N, Hanefeld M, Holt S, Jansky P, Keltai M, Lanas F, Leiter LA, Lopez-Jaramillo P, Cardona Munoz EG, Pirags V, Pogosova N, Raubenheimer PJ, Shaw JE, Sheu WH, Temelkova-Kurktschiev T; REWIND Investigators. Dulaglutide and cardiovascular outcomes in type 2 diabetes (REWIND): a double-blind, randomised placebo-controlled trial. Lancet. 2019 Jul 13;394(10193):121-130. doi: 10.1016/S0140-6736(19)31149-3. Epub 2019 Jun 9. PMID 31189511
- [Background] Pratley RE, Aroda VR, Lingvay I, Ludemann J, Andreassen C, Navarria A, Viljoen A; SUSTAIN 7 investigators. Semaglutide versus dulaglutide once weekly in patients with type 2 diabetes (SUSTAIN 7): a randomised, open-label, phase 3b trial. Lancet Diabetes Endocrinol. 2018 Apr;6(4):275-286. doi: 10.1016/S2213-8587(18)30024-X. Epub 2018 Feb 1. PMID 29397376
- [Background] Marso SP, Holst AG, Vilsboll T. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2017 Mar 2;376(9):891-2. doi: 10.1056/NEJMc1615712. No abstract available. PMID 28249135
- [Background] Wilding JPH, Batterham RL, Calanna S, Davies M, Van Gaal LF, Lingvay I, McGowan BM, Rosenstock J, Tran MTD, Wadden TA, Wharton S, Yokote K, Zeuthen N, Kushner RF; STEP 1 Study Group. Once-Weekly Semaglutide in Adults with Overweight or Obesity. N Engl J Med. 2021 Mar 18;384(11):989-1002. doi: 10.1056/NEJMoa2032183. Epub 2021 Feb 10. PMID 33567185
- [Background] Seijas-Amigo J, Salgado-Barreira A, Castelo-Dominguez R, Pereira-Pia M, Rodriguez-Manero M, Gonzalez-Juanatey JR. Semaglutide versus GLP-1 agonists. Effectiveness, safety, and quality of life in patients with diabetes mellitus 2. The SEVERAL study. Farm Hosp. 2022 Aug 30;46(6):372-379. PMID 36520578
- [Derived] Seijas-Amigo J, Salgado-Barreira A, Castelo-Dominguez R, Perez-Alvarez MT, Ponce-Pinon B, Fernandez-Silva M, Rodriguez-Barreiro M, Pereira-Pia M, Iglesias-Moreno JM, Gago-Garcia M, Montans-Garcia R, Fernandez-Perez A, Fraga-Gayoso D, Fernandez-Montenegro M, Riveiro-Barciela B, Rilla-Villar N, Cardeso-Paredes B, Ribeiro-Ferreiro M, Rodriguez-Penas D, Cordero A, Rodriguez-Manero M, Gonzalez-Juanatey JR; SEVERAL INVESTIGATORS. Effects of GLP-1 agonists on 10-year cardiovascular risk reduction in primary prevention: A 44-week open label prospective study. Diabetes Metab Syndr. 2025 Sep;19(9):103312. doi: 10.1016/j.dsx.2025.103312. Epub 2025 Oct 19. PMID 41129847
- See also: Dulaglutide datasheet — http://cima.aemps.es/cima/dochtml/ft/114956002/FT_114956002.html
- See also: Tofacitinib datasheet — http://cima.aemps.es/cima/dochtml/ft/114956002/FT_114956002.html
- See also: Exenatide datasheet — http://cima.aemps.es/cima/dochtml/ft/111696003/FT_111696003.html
- See also: Liraglutide datasheet — http://cima.aemps.es/cima/dochtml/ft/09529002/FT_09529002.html
- See also: Lixisenatide datasheet — http://cima.aemps.es/cima/dochtml/ft/12811005/FT_12811005.html
- See also: Semaglutide datasheet — http://cima.aemps.es/cima/dochtml/ft/117251002/FT_117251002.html